CLINICAL TRIAL: NCT02030171
Title: Effect of Three Therapeutic Strategies on the Restriction of the Participation of Patients With a Chronic Back Pain : Multidisciplinary is it the Key Component ?
Brief Title: Effect of Three Therapeutics Strategies on Patients With a Chronic Back Pain (PLURICLEF).
Acronym: PLURICLEF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49RC08_0014
Record Dates: First submitted 2013-12-19; First posted 2014-01-08 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic low back pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PLURIHOC (Active Comparator): -Functionnal reeducation : in hospital, intensive, multidisciplinary.
  Interventions: Other: functionnal reeducation
- KIPLURI (Active Comparator): -Functionnal reeducation : ambulatory, no intensive multidisciplinary.
  Interventions: Other: functionnal reeducation
- KIMONO (Active Comparator): -Functionnal reeducation : ambulatory, low-intensity
  Interventions: Other: functionnal reeducation

INTERVENTIONS:
Other: functionnal reeducation — Specific functionnal reeducation for chronic low back pain

SUMMARY:
Effect of three therapeutics strategies on the restriction of the participation of patients with a chronic back pain : multidisciplinary is it the key component ?

DETAILED DESCRIPTION:
Compare the efficacy of 1 year of participation, of three programs of care for patients with chronic law back, referred to specialists rehabilitation centers or directly to the multidisciplinary consultation of university hospital of Angers.

The primary objectif is to assess the efficacy of 1 year of the three therapeutics strategies with the number of days off work in the year following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Obtaining the signature of consent to participate in the study.
* Male or female, aged 18-55 years.
* Diagnosis of common chronic low back pain.
* Chronic low back pain that led to at least a month off work in the previous year or at least 3 months of stops in the previous 2 years.
* Employee and holds a permanent contract or a fixed-term contract in the public or private sector.

Exclusion Criteria:

* Lack of consent to participate in the study.
* No possibily to follow one of three programs of study
* Pregnant women, new mothers or mothers who are breastfeeding.
* No affiliation to the french social system.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2009-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Efficiency of the 3 programs | One year
  Compare the efficacy of 1 year of participation of the three programs of care for chronic low back pain patients referred to specialists rehabilitation centers or directly to the multidisciplinary consultation UH Angers.
  The primary endpoint to assess the efficacy of 1 year of support on the participation of the patient is the number of days off work in the year following treatment.

SECONDARY OUTCOMES:
Evolution of quality of life scales | One year
  The secondary endpoints to assess the efficacy of 1-year quality of life of the patient is the SF-36 score.
  The quality of life questionnaire is collected early in the program at the end (after the 5-week program ended) at 6 months and one year.
Compare the effectiveness of 1 year on improving the social integration of three programs supported in the same patients. | One year
  The secondary endpoint to assess the efficacy of 1 year of support on improving social inclusion is the score of Dallas.
  The Dallas questionnaire is collected early in the program at the end (after the 5-week program ended) at 6 months and one year.
Compare the effectiveness of 1 year on physical deconditioning, three programs of care in these patients. | One year
  The secondary endpoints to assess efficacy at 1 year of support on the physical deconditioning of the patient are the finger-floor distance, Ito test, and the test port heavy load.
  These tests are performed early in the program at the end (after the program ended five weeks) at 6 months and one year.
Compare the cost of 1 year from the point of view of health insurance, of the three therapeutic strategies. | One year
  The secondary endpoints to assess the cost of 1 year from the point of view of health insurance, are the direct and indirect costs.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Richard-Crémieux, Md-PhD, Principal Investigator — UH Angers
Locations (1):
- University Hospital of Angers, laboratory epidemiology, ergonomics and occupational health, Angers, Pays de Loire, France

REFERENCES:
- [Background] Bontoux L, Roquelaure Y, Billabert C, Dubus V, Sancho PO, Colin D, Brami L, Moisan S, Fanello S, Penneau-Fontbonne D, Richard I. [Prospective study of the outcome at one year of patients with chronic low back pain in a program of intensive functional restoration and ergonomic intervention. Factors predicting their return to work]. Ann Readapt Med Phys. 2004 Oct;47(8):563-72. doi: 10.1016/j.annrmp.2004.03.006. French. PMID 15465161
- [Background] Leclerc A, Chastang JF, Ozguler A, Ravaud JF. Chronic back problems among persons 30 to 64 years old in France. Spine (Phila Pa 1976). 2006 Feb 15;31(4):479-84. doi: 10.1097/01.brs.0000199939.53256.e0. PMID 16481962
- [Background] Leggett S, Mooney V, Matheson LN, Nelson B, Dreisinger T, Van Zytveld J, Vie L. Restorative exercise for clinical low back pain. A prospective two-center study with 1-year follow-up. Spine (Phila Pa 1976). 1999 May 1;24(9):889-98. doi: 10.1097/00007632-199905010-00010. PMID 10327511
- [Background] Jousset N, Fanello S, Bontoux L, Dubus V, Billabert C, Vielle B, Roquelaure Y, Penneau-Fontbonne D, Richard I. Effects of functional restoration versus 3 hours per week physical therapy: a randomized controlled study. Spine (Phila Pa 1976). 2004 Mar 1;29(5):487-93; discussion 494. doi: 10.1097/01.brs.0000102320.35490.43. PMID 15129059
- [Background] Biering-Sorensen F. Physical measurements as risk indicators for low-back trouble over a one-year period. Spine (Phila Pa 1976). 1984 Mar;9(2):106-19. doi: 10.1097/00007632-198403000-00002. PMID 6233709
- [Derived] Ronzi Y, Roche-Leboucher G, Begue C, Dubus V, Bontoux L, Roquelaure Y, Richard I, Petit A. Efficiency of three treatment strategies on occupational and quality of life impairments for chronic low back pain patients: is the multidisciplinary approach the key feature to success? Clin Rehabil. 2017 Oct;31(10):1364-1373. doi: 10.1177/0269215517691086. Epub 2017 Feb 13. PMID 28592147
- [Derived] Petit A, Roche-Leboucher G, Bontoux L, Dubus V, Ronzi Y, Roquelaure Y, Richard I. Effectiveness of three treatment strategies on occupational limitations and quality of life for patients with non-specific chronic low back pain: Is a multidisciplinary approach the key feature to success: study protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2014 Apr 16;15:131. doi: 10.1186/1471-2474-15-131. PMID 24739659